CLINICAL TRIAL: NCT04735926
Title: Randomised, Double-blind, Double-dummy, Multicentre Trial to Evaluate the Efficacy and Safety of Three Different Weekly Dosages of Calcifediol Versus Placebo in Subjects With Either Vitamin D Deficiency or Insufficiency.
Brief Title: Efficacy and Safety of Calcifediol vs Placebo in Subjects With Vitamin D Deficiency
Acronym: WORFEROL
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Faes Farma, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HIDR-0320/DR
Record Dates: First submitted 2021-01-29; First posted 2021-02-03 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Vitamin D Deficiency; Vitamin D Insufficiency
Keywords: Vitamin D deficiency; Hypovitaminosis D; Vitamin D Insufficiency
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Calcifediol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Group 1A (Placebo Comparator): Subjects corresponding to Cohort 1 (25-OH-D baseline level > 10 to < 20 ng/mL)
  Interventions: Other: Placebo
- Group 1B (Experimental): Subjects corresponding to Cohort 1 (25-OH-D baseline level > 10 to < 20 ng/mL)
  Interventions: Drug: Calcifediol 75mcg; Other: Placebo
- Group 1C (Experimental): Subjects corresponding to Cohort 1 (25-OH-D baseline level > 10 to < 20 ng/mL)
  Interventions: Drug: Calcifediol 100mcg; Other: Placebo
- Group 2A (Placebo Comparator): Subjects corresponding to Cohort 2 (25-OH-D baseline level ≤ 10 ng/mL)
  Interventions: Other: Placebo
- Group 2B (Experimental): Subjects corresponding to Cohort 2 (25-OH-D baseline level ≤ 10 ng/mL)
  Interventions: Drug: Calcifediol 100mcg; Other: Placebo
- Group 2C (Experimental): Subjects corresponding to Cohort 2 (25-OH-D baseline level ≤ 10 ng/mL)
  Interventions: Drug: Calcifediol 125mcg; Other: Placebo

INTERVENTIONS:
Drug: Calcifediol 75mcg — Soft gelatin capsule. Oral administration once per week
  Arms: Group 1B
Drug: Calcifediol 100mcg — Soft gelatin capsule. Oral administration once per week
  Arms: Group 1C; Group 2B
Drug: Calcifediol 125mcg — Soft gelatin capsule. Oral administration once per week.
  Arms: Group 2C
Other: Placebo — Soft gelatin capsule. Oral administration once per week.
Other: Placebo — Soft gelatin capsule. Oral administration once per week.
  Arms: Group 1A; Group 2A

SUMMARY:
This is a randomised, double-blind, double-dummy, multicentre, dose-ranging clinical trial in subjects with vitamin D deficiency or insufficiency. Its general objective is to determine the efficacy and safety of different doses of calcifediol soft gelatin capsules (SGCs) compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects ≥ 18 years of age.
* Evidence of serum 25-OH-D levels < 20 ng/mL or ≤ 10 ng/mL, for each cohort.
* Written informed consent.
* For females of childbearing potential only: willing to perform pregnancy tests, must agree to use highly effective methods of birth control throughout the study.

Exclusion Criteria:

* Subjects receiving any treatment with calcifediol, vitamin D analogues, vitamin complexes or vitamin D supplements.
* Subjects taking drugs that could modify vitamin D levels.
* Subjects taking calcium supplements.
* Uncorrected hypercalcaemia, known hypercalciuria or nephrolithiasis.
* Severe renal impairment.
* Subjects diagnosed with liver or biliary failure, congestive heart failure, malabsorption, primary hyperparathyroidism, hypothyroidism, prolonged immobilisation, sarcoidosis, tuberculosis or other granulomatous diseases or hyperthyroidism.
* Any present or previous malignancy.
* Known contraindications or sensitivities to the use of the IP or any of its components.
* Pregnant woman, breastfeeding woman or woman planning a pregnancy.
* Subject has received an IP within 30 days before the start of the screening or is currently enrolled in an investigational interventional study.
* Any condition that may jeopardise the clinical trial conduct according to the protocol.
* Employees of the investigator or clinical trial site, as well as family members of the employees or the principal investigator.
* Person committed to an institution by virtue of an order issued either by judicial or other authorities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 674 (Actual)
Dates: Start 2020-12-23 (Actual); Primary Completion 2022-07-21 (Actual); Study Completion 2023-04-25 (Actual)

PRIMARY OUTCOMES:
To assess efficacy for each cohort in terms of percentage of subjects achieving 25-OH-D levels ≥ 30 ng/mL and/or ≥ 20 ng/mL at 16 weeks of treatment. | 16 weeks
  Percentage of subjects who achieve 25-OH-D levels ≥ 30 ng/mL and/or ≥ 20 ng/mL

CONTACTS AND LOCATIONS:
Locations (55):
- Bulgaria (7):
  - MC-1-Sevlievo Ltd., Sevlievo
  - Diagnostic & Consultative Center "Sveta Anna" EOOD, Sofia
  - Individual Practice Ambulatory for Specialized Medical Care - Cardiology, Obstetrics and Gynecology, Sofia
  - IV MHAT - Sofia, Sofia
  - Lora - Medical center Sofia, Sofia
  - Medical Centre Asklepion - Research in human medicine, Sofia
  - Medical Centre Salvebis, Sofia
- Czechia (11):
  - Alergologie Němcová, s.r.o., Brno
  - Poliklinika Choceň - Neurologická ambulance, Choceň
  - MUDr. Eva Richterová - HK, s.r.o., Hradec Králové
  - MUDr. Tomáš Edelsberger, Krnov
  - G-CENTRUM Olomouc s.r.o., Olomouc
  - Centrum gynekologické rehabilitace s.r.o., Písek
  - Centrum pro diagnostiku a léčbu myasthenia gravis - Neurologická klinika 1. LF UK a VFN v Praze, Prague
  - MediCel, s.r.o., Prague
  - Milan Kvapil s.r.o., Prague
  - RS centrum - Neurologická klinika 1.LF UK a VFN v Praze, Prague
  - Ordinace MediFem, s.r.o., Teplice
- France (4):
  - CHU Bordeaux, Hôpital Pellegrin, Bordeaux
  - CHR Orléans, Service Rhumatologie, Orléans
  - CHU Saint Etienne, Hôpital Nord, Saint-Etienne
  - CHU Purpan, Toulouse
- Italy (6):
  - Fondazione IRCCS Cà Granda - Ospedale Maggiore Policlinico -UOC Endocrinologia e Malattie Metaboliche, Milan
  - IRCCS Ospedale San Raffaele /Unità di Endocrinologia, Milan
  - Azienda Ospedaliero Universitaria - Università degli Studi della Campania Luigi Vanvitelli - UOC di Medicina Fisica e Riabilitazione, Napoli
  - UOC di Riabilitazione -Azienda Ospedaliero Universitaria Paolo Giaccone Palermo, Palermo
  - AOU Pisana - Centro di Farmacologia Clinica per la Sperimentazione dei Farmaci, Pisa
  - Fondazione PTV -Policlinico Ospedaliero Universitario Tor Vergata - U.O.C. Ortopedia e Traumatologia, Roma
- Serbia (6):
  - Institut za reumatologiju, Belgrade
  - Klinički centar Kragujevac, Centar za reumatologiju, alergologiju i kliničku imunologiju, Odeljenje za reumatologiju, Kragujevac
  - Institut za lečenje i rehabilitaciju "Niška Banja" Niš, Klinika za reumatologiju, Niška Banja
  - Klinički centar Vojvodine, Klinika za endokrinologiju, dijabetes i bolesti metabolizma, Novi Sad
  - Specijalna bolnica za reumatske bolesti Novi Sad, Novi Sad
  - Opšta bolnica "Đorđe Joanović" Zrenjanin, Odeljenje za reumatologiju, Zrenjanin
- Slovakia (13):
  - IN MEDIC s.r.o., Neurologická ambulancia, Bardejov
  - ALERGO H2B, s.r.o., Ambulancia klinickej imunológie a alergológie, Komárno
  - ALERSA, s.r.o., Ambulancia klinickej imunológie a alergológie, Košice
  - Endomed, s.r.o. - Gastroenterologická ambulancia, Košice
  - DANIMED, s.r.o., Ambulancia klinickej imunológie a alergológie, Levice
  - KARDIO 1, s.r.o., Kardiologická ambulancia, Lučenec
  - Elte HU, s.r.o., Chirurgická ambulancia, Rimavská Sobota
  - Kardioamb, s.r.o., Kardiologická a interná ambulancia, Rimavská Sobota
  - MEDILEX, s.r.o., Ambulancia vnútorného lekárstva, Rimavská Sobota
  - Zoll-Med, s.r.o., Ambulancia klinickej imunológie a alergológie, Rimavská Sobota
  - Pľúcna ambulancia Hrebenár, s.r.o. - Pneumologicko-ftizeologická ambulancia, Spišská Nová Ves
  - ANA JJ, s.r.o., Ambulancia klinickej imunológie a alergológie, Topoľčany
  - KK Neuro, s.r.o., Neurologická ambulancia, Žilina
- Spain (8):
  - Clínica Sagrada Familia, Barcelona
  - EAP Sardenya, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Quirónsalud Barcelona, Barcelona
  - Hospital Universitario Quirónsalud Madrid, Pozuelo de Alarcón
  - Complejo Asistencial Universitario de Salamanca, Salamanca
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Universitario Rio Hortega, Valladolid

IPD SHARING:
Plan to Share IPD: No